CLINICAL TRIAL: NCT02583529
Title: Neurogenic Overactive Bladder Treatment on Parkinson's Disease Through Back Tibial Nerve Electrostimulation
Acronym: NOVTPD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tatiane Gomes de Araujo (Other)
Responsible Party: Sponsor-Investigator, Tatiane Gomes de Araujo, MD, Hospital de Clinicas de Porto Alegre
Organization: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0554
Record Dates: First submitted 2015-09-26; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Overactive Bladder; Parkinson Disease
Keywords: Parkinson Disease; Neurogenic Overactive Bladder; Posterior Tibial Nerve Electrostimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Back Tibial Nerve Electrostimulation (Experimental): They will be assessed before and after 12 weeks of treatment with home PTNE through specific form of questionnaires assessing incontinence, quality of life and voiding diary. After the end of treatment will be made up of patients to verify the effectiveness of treatment in 30 to 90 days.
  Interventions: Device: Back Tibial Nerve Electrostimulation
- Placebo Electrostimulation (Placebo Comparator): They will be assessed before and after 12 weeks of treatment with home PTNE through specific form of questionnaires assessing incontinence, quality of life and voiding diary. After the end of treatment will be made up of patients to verify the effectiveness of treatment in 30 to 90 days.
  Interventions: Device: Placebo Electrostimulation

INTERVENTIONS:
Device: Back Tibial Nerve Electrostimulation — The BTNE will be made with electrodes Silver Spike Point (SSP) set in an ankle with the negative pole positioned on the inner malleolus and the positive approximately 05 cm below the previous, and connected to a portable stimulator powered by rechargeable battery developed by the Biomedical Engineering Department of the HCPA.
  Arms: Back Tibial Nerve Electrostimulation
Device: Placebo Electrostimulation — The BTNPE will be made with electrodes Silver Spike Point (SSP) set in an ankle with the negative pole positioned on the inner malleolus and the positive approximately 05 cm below the previous, and connected to a portable stimulator powered by rechargeable battery developed by the Biomedical Engineering Department of the HCPA.
  Arms: Placebo Electrostimulation

SUMMARY:
Dysfunctions of the lower urinary tract are non-motor symptoms common engines in Parkinson's disease (PD). Urodynamic changes in PD include overactive bladder (OB), characterized by urgency with or without urge incontinence , usually with frequency and nocturia . The aim of this study is to evaluate the efficacy and effectiveness of the treatment of OB in patients with PD with the use of a specific treatment: Posterior Tibial Nerve Electrostimulation (PTNE).

DETAILED DESCRIPTION:
Introduction: Dysfunctions of the lower urinary tract are non-motor symptoms common engines in Parkinson's disease (PD). Urodynamic changes in PD include overactive bladder (OB), characterized by urgency with or without urge incontinence , usually with frequency and nocturia . The aim of this study is to evaluate the efficacy and effectiveness of the treatment of OB in patients with PD with the use of a specific treatment: Posterior Tibial Nerve Electrostimulation (PTNE). Materials and methods: This is test-clinical, double-blind, randomized, controlled comparison with placebo. The research will be conducted with patients diagnosed with PD and symptoms of OB in the Clinical Hospital of Porto Alegre, in the Movement Disorders and Urogynecology Ambulatories. The patients are divided into two groups, one of which receives placebo stimulation (often below the therapeutic threshold). They will be assessed before and after 12 weeks of treatment with home PTNE through specific form of questionnaires assessing incontinence, quality of life and voiding diary. After the end of treatment will be made up of patients to verify the effectiveness of treatment in 30 to 90 days. Hypothesis: Through this research the investigators hope to determine the true efficacy of this treatment method with PTNE in OB in PD with a high level of evidence, seeking to improve urinary symptoms and quality of life in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD according to the criteria of the London Brain Bank
* Complaint urinary storage symptoms such as urinary urgency (sudden urge, abrupt and imperious to urinate, which is difficult to be inhibited), with or without urge incontinence (urine leakage after emergency), frequency (number of urination> 7 / day) and nocturia (the number of micturitions> 1 / night).

Exclusion Criteria:

* Damage to the peripheral sacral nerves
* Infection of the lower urinary tract untreated;
* Diabetes Mellitus;
* Chronic pulmonary disease worsened;
* Pregnancy and postpartum;
* Urinary Incontinence of pure stress incontinence or urinary Mixed with predominance of the stress component;
* Pacemaker or defibrillator;
* Metal prostheses;
* Application of botulinum toxin into the bladder and / or pelvic muscles last year;
* Current TENS treatment in the pelvic region, lower back and / or legs;
* Prior Urinary incontinence surgery;
* Current bladder carcinoma;
* Cognitive impairment likely to prevent implementation of the proposed treatment;
* Not understand / sign informed consent.

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Voiding diary | 3 months
  Consists of daily annotation fluid intake, frequency (number) and volume of urination (mL), daily activities and episodes of incontinence (number), need and number of hygienic protections, etc. It is a cost-effective method of initially assessing urinary complaints when compared to the test pad (pad test) and standardized symptom scales.The voiding diary will be filled before and after treatment that will last 03 months (baseline and 3 months). The patient will record your urinary habits for one day (24 hours) before starting treatment and after completion.

SECONDARY OUTCOMES:
Hoehn and Yahr Disability Stage of scale | 3 months
  Developed in 1967, called the DP indication of the general state of the patient. It comprises five phases (Table 1). On this scale, patients classified in stages 1, 2 and 3 show mild to moderate disability, while in stages 4 and 5 show more severe disability. HY is applied before treatment (baseline).
King's Health Questionnaire | 3 months
  The questionnaire presents 32 items distributed into 10 domains and is available in 26 languages. A change from baseline of 5 points (out of 100) in any field indicates significant clinical improvement. KHQ is applied before and after treatment (baseline and 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Geraldo Lopes Ramos, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Tatiane Gomes de Araujo, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Araujo TG, Schmidt AP, Sanches PRS, Silva Junior DP, Rieder CRM, Ramos JGL. Transcutaneous tibial nerve home stimulation for overactive bladder in women with Parkinson's disease: A randomized clinical trial. Neurourol Urodyn. 2021 Jan;40(1):538-548. doi: 10.1002/nau.24595. Epub 2020 Dec 16. PMID 33326648